CLINICAL TRIAL: NCT01725997
Title: Operative or Conservative Treatment of Acute Acromioclavicular Joint Dislocation Rockwood Grade III and V - a Prospective Randomized Study
Brief Title: Operative or Conservative Treatment of Acute Acromioclavicular Joint Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Goran's Hospital (Other)
Responsible Party: Principal Investigator, Helena Boström Windhamre, MD, St Goran's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC-lux
Record Dates: First submitted 2012-10-31; First posted 2012-11-14 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Acromioclavicular Joint Dislocation
Keywords: acromioclavicular joint dislocation; ac joint dislocation; acromioclavicular joint separation; hook plate; Rockwood
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative treatment (Active Comparator): Operative treatment with hook plate.
  Interventions: Procedure: hook plate
- Conservative treatment (Active Comparator): Physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Procedure: hook plate — Surgery with hook plate followed by physiotherapy
  Other Names: hook plate by Synthes
  Arms: Operative treatment
Other: Physiotherapy — Patients will be following a program specific for AC joint dislocations
  Arms: Conservative treatment

SUMMARY:
The study aims to answer if surgery with hook plate for acute dislocation of the acromioclavicular joint (AC joint) grade III and V according to Rockwood is superior to conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* AC joint dislocation grade III according to Rockwood with at least half a clavicular bone width above the acromion or grade V according to Rockwood
* men and women 18-65 years and able to work
* understand spoken and/or written Swedish or English language
* be able to start treatment within 3 weeks from trauma
* consent form signed

Exclusion Criteria:

* earlier injury to, or surgery of either of the shoulders
* simultaneous fracture of the clavicle or acromion
* associates neurovascular injury
* severe osteoporosis
* open dislocation
* open growth plate of the acromion
* local skin damage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Constant Score | change from Baseline in Constant Score at 24 months

SECONDARY OUTCOMES:
Disabilities of Arm, Shoulder and Hand function (QuickDASH) | change from Baseline in QuickDASH at 24 months

OTHER OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Change from baseline in SPADI at 24 months
Radiographs with and without weight | Change in the position of the AC-joint from baseline to at 24 months
  Position of the AC-joint will be measured at standard radiographs and weighted radiographs
European Quality of Life - 5 dimensions (EQ5D) | Change from baseline in EQ-5D at 24 months
Pain rated with Visual Analogue Scale (VAS) | Change from baseline in VAS at 24 months
Computed Tomography | Change in the position of the AC-joint from baseline to at 24 months
  Position of the AC-joint

CONTACTS AND LOCATIONS:
Overall Officials: Helena Boström Windhamre, Principal Investigator — Capio St Gorans hospital
Locations (1):
- Capio St Gorans Hospital AB, Stockholm, Sweden